CLINICAL TRIAL: NCT04971083
Title: Intervention Phase: Patient-centered Nutrition Care (PaCC II)
Brief Title: Patient-centered Nutrition Care II: An E-health Supported Symptom Based Nutrition Intervention
Acronym: PaCC II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Cankado GmbH (Industry)
Responsible Party: Principal Investigator, PD Dr. med. Volker Heinemann, Professor Doktor, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PaCC II
Record Dates: First submitted 2021-06-24; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Nutritional Status; Psychological Distress; Quality of Life; Weight Change, Body
MeSH Terms: conditions — Body Weight Changes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Control (CG): receives Usual Care. Observational data regarding energy and fluid intake, weight, quality of life, symptoms, and distress status will be recorded in the Electronic Health Platform. They will have to ability to print and share this documentation with their HCP at their own discretion.
  Inflammation status will be recorded when data from routine blood draws is available
- Intervention Group (Active Comparator): Intervention Group (IG): The intervention consists of a built-in automated analysis that provide patient-tailored nutrition recommendations and behavioural tipps. Described in detail this means that dependent on the severity of the nutrition related symptom burden (NRSB) recorded, the patients in the intervention group only are, for example provided with detailed written nutrition information and cooking recipes and/or asked to discuss the symptoms with their health care provider, dietitian, and/or physician, or even asked to seek immediate medical care.
  Analog to the control group, observational data regarding energy and fluid intake, weight, quality of life, symptoms, and distress status will be recorded in the Electronic Health Platform. They will have to ability to print and share this documentation with their HCP at their own discretion.
  Inflammation status will be recorded when data from routine blood draws is available
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — This study is designed to provide patients a tool with which they can record the nutrition related symptom burden (NRSB) they are experiencing in real time. A pre-defined algorithm then provides them with tailored nutrition information and behavioural tipps based on the severity grade of the symptom recorded. The aim is to increase the chances that such symptoms, when clinically relevant, are addressed in a timely matter and thus the nutrition status is stabilized.
  Other Names: Electronic health information platform with active behavioural tipps
  Arms: Intervention Group

SUMMARY:
The aim of this study is to utilize the E-Health platform (EHIP) containing behavioural tipps to enable the provision of early appropriate nutrition recommendations to patients undergoing cancer therapy thereby stabilizing the nutrition status as measured with the scored Patient-Generated Subjective Global Assessment. Furthermore, we plan to explore the causal pathway between the change in the number and severity of nutrition related symptoms, measure the difference in weight change in percent between the two groups, determine a change in the level of the distress status, and measure the change in functional status. This Information could provide a basis for future nutrition intervention strategies aimed at improving overall nutrition status of patients undergoing cancer therapy and could potentially improve clinical and functional outcomes of this population.

DETAILED DESCRIPTION:
Primary Endpoint:

Nutrition care, augmented with E-Health tools containing tailored behavioural tipps enable the maintenance of overall nutrition status 12 weeks from baseline as measured with the Scored Patient-Generated Subjective Global Assessment. .

Secondary Endpoints will include:

* difference in the two arms in % weight loss
* difference in the number and severity of further Patient Reported nutrition relation symptoms according to Patient Reported- Common Toxicity Criteria for adverse events (PRO-CTCAE™) developed by the Division of Cancer Control and Population Sciences in the National Cancer Institute Version date: 2/25/2019
* change in Quality of Life as measured by Functional Assessment of Cancer Therapy - General questionnaire
* improvement of nutrition status
* change in the % of estimated energy intake achieved
* difference of the number of discontinuations or delay in therapy
* difference of Glasgow Prognostic Score (only when C-reactive protein und Albumin are available in the routine blood draw)
* change in Distress status

Study Design:

This mono-centric prospective randomized study is designed to test the hypothesis of a causal pathway between nutritional interventions containing tailored behavioural tipps augmented with E-health tools on predefined outcomes (nutrition status, weight loss, extent and severity of nutrition related symptom burden (NRSB), distress status QoL) The study will utilize E-Health tools to ensure regular and early identification of potential nutrition related symptoms on the part of both the patient and the clinician. Within this framework, the trial will include cancer patients with tumors in the GI tract undergoing chemo and/or immune therapy who will receive therapy for a minimum of six weeks after recruitment.

Study Methods:

Control (CG): receives Usual Care (Nutrition intervention according to house standards: Nutrition Risk Score ≥ 3, or patient, or clinician request). Additionally, patients will record their energy intake, weight, general state of being, symptoms, and distress status in the Electronic Health Platform (EHIP) and have to ability to print and share this documentation with their health care providers (HCP) at their own discretion.

Intervention Group (IG): analog to the control group, patients record their energy intake, weight, general state of being, symptoms, and distress status in the Electronic Health Platform (EHIP). A built-in automated analysis will provide patient-tailored nutrition recommendations. Dependent on the severity of the NRSB recorded, they are, for example, provided with detailed written nutrition information and cooking recipes aimed at and/or asked to discuss their symptoms with their dietitian, physician, or, if necessary, to seek immediate medical care. As in the control group, patients will also have the ability to print and share this documentation with their HCP at their own discretion.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients with tumors in the GI tract undergoing chemo and/or Immunotherapy and are primarily treated on an outpatient basis
* ≥ 18 years
* Life expectancy ≥ 6 months
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
* Open for, and ability to use, of E-Health platforms (own and uses one or more electronic devices with access to internet)
* Able to take 75% of foods orally
* Valid declaration of consent to participate in the study

Exclusion Criteria:

* Cancer patients with other diagnoses or who are not receiving chemo or Immunotherapy or undergoing intensive therapy requiring longer in-patient stays (e.g: Intensive Care Patients)
* ≤ 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≥3
* More than 75% of Energy intake is not taken oral but instead via enteral or parenteral route.
* Operation planned during the course of the Study (next 3 months)
* Patient who do provide not or withdraw their consent
* Not open or willing to use E-Health tools

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12-28 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Stabilization of patient-reported nutrition nutrition status | 12 weeks from baseline
  A automated analysis embedded in the E-health tool will provide patient-tailored nutrition information and behavior advice aimed at stabilizing or improving nutrition status. Nutrition status will be measured using the scored Patient-Generated Subjective Global Assessment (scale of 1-36) whereas a higher score indicates a declining nutrition status

SECONDARY OUTCOMES:
Number and severity of patient-reported nutrition related symptoms between the groups | 12 weeks from baseline
  Difference of the number and severity of patient-reported nutrition related symptoms according to Patient Reported- Common Toxicity Criteria for adverse events (PRO-CTCAE™) developed by the Division of Cancer Control and Population Sciences in the National Cancer Institute Version date: 2/25/2019. 13 Symptoms will be measured for frequency and severity.
Weight change | 12 weeks from baseline
  Difference in percent of weight change between the groups
Quality of life improvement | 12 weeks from baseline
  Improvement of Quality of life as measured by the Functional Assessment of Cancer Therapy - General (FAKT-G) questionnaire. According the scale of 0-108 the higher the score, the better the QOL.
Improvement of nutrition intake | 12 weeks from baseline
  % of estimated energy intake
Discontinuations or delay in therapy reduction | 12 weeks from baseline
  no. of discontinuations or delay in therapy
Inflammation status | 12 weeks from baseline
  change in Glasgow Prognostic Score on a scale of 0-2 (only when C-reactive Protein und Albumin are available in the routine blood draw). A higher score indicates more inflammation
Distress status | 12 weeks from baseline
  change in Distress state measured by Distress Thermometer on a scale of 1-10. A higher the score indicates more Distress

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Erickson, M.Sc., Principal Investigator — CCC Ludwig Maximillian University Munich; Julian Holch, PD, MD, Principal Investigator — CCC Ludwig Maximillian University Munich
Locations (1):
- Comprehensive Cancer Center Ludwig Maximilian University Munich, Munich, Barvaria, Germany

IPD SHARING:
Plan to Share IPD: No